CLINICAL TRIAL: NCT06930976
Title: Tracing Of Real-time glu13Cose Metabolism in Human Immune Cells
Acronym: TORCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Stier, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 241348
Record Dates: First submitted 2025-04-08; First posted 2025-04-16 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Glucose; Metabolism; Isotope Labeling; Immune System and Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 13C6-Glucose (Other): 10-25gm of 13C6-Glucose
  Interventions: Drug: 13C6-Glucose

INTERVENTIONS:
Drug: 13C6-Glucose — Compounded as 5% 13C6-Glucose in sterile water given IV over 2-4 hours as a split bolus and infusion

SUMMARY:
The purpose of this study is to understand how cells of the immune system use the common sugar glucose to fuel energy production and as a building block within the cell. Investigators will intravenously infuse a non-radioactive glucose tracer into participants over a few hours and collect immune cells from the blood to track uptake and usage of this glucose within these immune cells.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older

Exclusion Criteria:

* Pregnant
* Prisoner or in police custody
* Uncontrolled hyperglycemia/diabetes
* Current participation in another study where the total volume of blood drawn, when added to this study blood draw volume, exceeds 500cc in an 8 week period
* Any medical issue or pharmacologic exposure which, in the opinion of the study investigator, that might interfere with the study objectives
* Any reason which, in the opinion of the study investigator, adds additional risk to the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
13C6-glucose uptake in immune cells | Up to 4 hours
  Detection of 13C6-glucose-derived metabolites in neutrophils, monocytes, CD4 T cells, and CD8 T cells using gas and liquid chromatography-mass spectrometry (GC-MS and LC-MS) following magnetic enrichment of these immune cell subsets.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T Stier, M.D., Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available after de-identification.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will become available within 6 months of publication of the outcomes and will remain available for at least 5 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Principle Investigator and relevant institutional review boards.